CLINICAL TRIAL: NCT01952860
Title: A Feasibility Study of Hatha Yoga in Couples Coping With Lung Cancer
Brief Title: Hatha Yoga in Lung Cancer Couples
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Requested by PI during yearly Continuing Review
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0496
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Non-small cell lung cancer; NSCLC; Caregiving partner; Hatha Yoga; Radiation therapy; XRT; Questionnaires; Surveys
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hatha Yoga (Experimental): Participants receive 18 sessions of Hatha yoga over the course of radiation therapy. Each 45 to 60 minute session guided by an instructor. Participant should attend each session together with their caregiving partner. Some sessions videotaped. At first session, participant given a CD and instructions for practicing Hatha yoga at home. Questionnaire completion at baseline, during radiation therapy, and at completion of radiation therapy.
  Interventions: Other: Hatha Yoga; Behavioral: Questionnaires

INTERVENTIONS:
Other: Hatha Yoga — 18 sessions of Hatha yoga over the course of radiation therapy. Each 45 to 60 minute session guided by an instructor. Participant should attend each session together with their caregiving partner. Some sessions videotaped. At first session, participant given a CD and instructions for practicing Hatha yoga at home.
Behavioral: Questionnaires — Questionnaire completion at baseline, during radiation therapy, and at completion of radiation therapy.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn the opinion of patients and their caregiving about a couple-based Hatha Yoga program during treatment for cancer. Researchers also want to learn the effect of this program on lung function, distress, and quality of life.

DETAILED DESCRIPTION:
If participant agrees to take part, participant's medical history and demographic information (such as age, sex, and race) will be recorded. By signing this consent, participant also agrees that participant's caregiving partner will be approached to take part in this study.

Questionnaires:

Participant will complete about 10 questionnaires before participant's first radiation treatment and again after participant completes participant's treatment schedule (usually 6 weeks later). The questionnaires ask about participant's health, any symptoms participant may be having, participant's mood, participant's level of fatigue, participant's sleeping habits, participant's relationship, and participant's quality of life. It should take about 45 minutes to complete these questionnaires.

Participant will complete about 5 questionnaires again halfway through participant's radiation treatment schedule. These questionnaires ask about participant's quality of life. These should take about 20 minutes to complete.

During each week of radiation therapy, participant will also complete a questionnaire asking participant's feelings about the Hatha Yoga sessions. Participant will be asked to list what participant liked or disliked, what participant found most and least useful, and how participant would rate the instructor. Participant will also be asked about how often participant practices outside of class and if participant thinks they are benefitting from the Hatha Yoga program. It should take about 5 minutes to answer this questionnaire. Participant's answers to the questions will not be shared with participant's caregiving partner.

Hatha Yoga Sessions:

Participant will take part in up to 18 sessions of Hatha yoga over the course of radiation therapy. Each 45- to 60-minute session will be guided by an instructor. Participant should attend each session together as a couple.

During the yoga sessions, participant will be asked to do deep-breathing exercises and perform different stretching and movement exercises. The movements are designed not to be difficult, and participant will sit on the floor or in a chair while participant does them. Participant can move through the exercises at participant's own pace. The instructor will be available to answer any questions participant may have about the practice of Hatha yoga. Most of the yoga sessions may be videotaped. This is so the researchers can keep track of the quality of the sessions. Only the study staff will be able to view this videotape. The video files are digital and will be deleted after all the data are studied.

At participant's first session, participant will be given a CD and instructions for practicing Hatha yoga at home. While participant is receiving radiation therapy, participant will be asked to practice at home 1 time a day either with participant's caregiving partner or alone on the days participant does not have a session at the clinic.

Length of Study:

Participation on this study will be over when participant has completed the questionnaires during participant's last week of radiation therapy.

This is an investigational study.

Up to 15 patients and their caregiving partners, for a total of 30 participants, will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-small cell lung cancer (NSCLC) stages I through IIIB who are going to receive at least 5 weeks of thoracic radiation therapy with or without chemotherapy undergoing daily radiation treatment in the Department of Radiation Oncology at M. D. Anderson Cancer Center (MDACC) and an eligible and consenting caregiving partner.
2. Patients and caregiving partners must both be at least 18 years old.
3. Participants have a study eligible and consenting caregiving partner spouse or significant other (e.g, romantic partner). (i.e. spouse, romantic/domestic partners, significant others).
4. Patients and caregiving partners should be able to read, write, and speak English.

Exclusion Criteria:

1. Patients who are not oriented to time, place, and person.
2. Patients who have practiced Tibetan or Hatha yoga in the year prior to diagnosis on a regular basis.
3. Lung cancer patients with a life expectancy of less than 6 months per attending physician estimation.
4. Lung cancer patients with the attending physician-rated Eastern Cooperative Oncology Group (ECOG) performance status score of greater than 2 at the time of radiotherapy initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-09-23 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of Yoga Program in Lung Cancer Participants Receiving Radiation determined by attendance | 6 weeks
  If over 50% of eligible participants participate and at least 80% of the participants are evaluable for follow-up (completing at least one follow-up assessment in the middle of radiotherapy and during the last week of radiotherapy), the study will be deemed feasible.
Feasibility of Yoga Program in Lung Cancer Participants Receiving Radiation determined by questionnaire responses. | 6 weeks
  If over 50% of eligible participants participate and at least 80% of the participants are evaluable for follow-up (completing at least one follow-up assessment in the middle of radiotherapy and during the last week of radiotherapy), the study will be deemed feasible.
  European Organization for Research and Treatment of Cancer (EORTC) Lung Cancer-specific Quality of Life Questionnaire (QLQ-LC13) used for the follow-up assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, PHD, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org